CLINICAL TRIAL: NCT03080324
Title: Sublingual Versus Endovenous Fentanyl for Pain Treatment in Trauma Patients in the ER - a Double-blind Randomized Prospective Study
Brief Title: Sublingual Versus Endovenous Fentanyl for Pain Treatment in Trauma Patients in the Emergency Room
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Sanitaria dell'Alto Adige (Other)
Responsible Party: Principal Investigator, Elisabeth Gruber, MD, Azienda Sanitaria dell'Alto Adige
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SABES 1
Record Dates: First submitted 2016-12-04; First posted 2017-03-15 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Acute Pain Due to Trauma
Keywords: Fentanyl; Transmucosal administration; Endovenous administration; Pain therapy
MeSH Terms: conditions — Agnosia | interventions — Fentanyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl sublingual + Placebo ev (Experimental): Fentanyl 100 µg sublingual in acute sever pain + NaCl 0,9% endovenous to mimic fentanyl ev
  Interventions: Drug: Fentanyl sublingual; Drug: Placebo ev
- Fentanyl ev + Placebo sublingual (Active Comparator): Fentanyl ev in acute sever pain + Sugar pill manufactured to mimic fentanyl sublingual
  Interventions: Drug: Fentanyl ev; Drug: Placebo sublingual

INTERVENTIONS:
Drug: Fentanyl sublingual — Fentanyl sublingual
  Other Names: Abstral
  Arms: Fentanyl sublingual + Placebo ev
Drug: Fentanyl ev — Fentanyl ev
  Other Names: Fentanest
  Arms: Fentanyl ev + Placebo sublingual
Drug: Placebo sublingual — Placebo sublingual
  Other Names: Placebo
  Arms: Fentanyl ev + Placebo sublingual
Drug: Placebo ev — Saline
  Other Names: Saline
  Arms: Fentanyl sublingual + Placebo ev

SUMMARY:
The purpose of this study is to determine the non-inferiority of the efficacy of sublingual given fentanyl versus endovenous given fentanyl for patients in the emergency departement.

DETAILED DESCRIPTION:
Fentanyl endovenous (ev) is an excellent analgesic drug for pain relief in acute traumatic pain. Fentanyl sublingual (Abstral ®) is an excellent analgesic drug in the breakthrough pain relief in oncologic patients.

The immediate (10 minutes) effect and the ease of administration of sublingual fentanyl could be a possibility for a fast pain relief in remote areas such as mountain rescue missions.

Patients will be recruited according to a randomized list to fentanyl ev or fentanyl sublingual versus placebo oral or placebo ev.

Safety issues like control of vital signs will be warranted

ELIGIBILITY:
Inclusion Criteria:

* Trauma on the limbs with a pain score of 4 or more
* ASA I - II

Exclusion Criteria:

* children < 18 years
* cognitive impairment: brain injury, intoxication, analgesia
* weight under 50 kg and more then 100 kg
* other injuries like chest trauma with respiratory insufficiency, suspect liver or spleen injury, amputation;
* chronic analgesic use or misuse
* allergy
* fear of needles
* pregnancy
* speech difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Pain - Relief | 1 hour
  Pain - Relief of 2 points on a 11 items pain scale (0 = non pain; 10 = unbearable pain)

SECONDARY OUTCOMES:
Practicability / handling of the two dosage forms of fentanyl in emergencies | 1 hour
  Practicability / handling
Patient comfort | 1 hour
  5 items Labert Scale
Adverse drug effects | 1 hour
  such as pruritus, nausea, dizziness
SpO2 (%) | 1 hour
  SpO2 < 92%

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Gruber, MG MSc, Principal Investigator — Südtiroeler Sanitätsbetrieb
Locations (1):
- Emergency Room of Bruneck Regional Hospital, Bruneck, Italy

IPD SHARING:
Plan to Share IPD: No